CLINICAL TRIAL: NCT01065038
Title: A Single Blind, Multi-centre, Randomised Multinational Phase III Study to Compare the Efficacy and Tolerability of Anagrelide vs Hydroxyurea in Patients With Essential Thrombocythaemia
Brief Title: Anagrelide vs. Hydroxyurea - Efficacy and Tolerability Study in Patients With Essential Thrombocythaemia
Acronym: ANAHYDRET
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AOP Orphan Pharmaceuticals AG (Industry)
Other Study IDs: AOP03007
Record Dates: First submitted 2010-02-08; First posted 2010-02-09 (Estimated); Last update posted 2010-10-06 (Estimated); Status verified 2005-09

CONDITIONS: Essential Thrombocythaemia
MeSH Terms: conditions — Thrombocythemia, Essential | interventions — anagrelide; Hydroxyurea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Anagrelide (Experimental)
  Interventions: Drug: Anagrelide
- Hydroxyurea (Active Comparator)
  Interventions: Drug: Hydroxyurea

INTERVENTIONS:
Drug: Anagrelide
  Arms: Anagrelide
Drug: Hydroxyurea
  Arms: Hydroxyurea

SUMMARY:
Study AOP 03-007 was designed as a pivotal study to test, if Anagrelide (Thromboreductin®)was not inferior to HU with respect to efficacy in patients with ET. This approach to demonstrate non-inferiority was based on the following decision points:

• ET is a rare disease and recruitment of large patient number (> 1600) to prove superiority was not considered possible.

. It was decided to recruit only treatment naïve high risk patients to avoid pre-treatment bias, which further limited the number of patients eligible for the study.

ELIGIBILITY:
Inclusion Criteria:

* Presence of essential thrombocythaemia with high-risk profile.

Exclusion Criteria:

* previous treatment with cytoreductive drugs or Anagrelide
* pregnant women or women in childbearing age with inadequate contraception
* patients with contraindications for study drugs due to anaphylactoid reactions to either active or non-active ingredients
* known lactose intolerance
* cardiovascular diseases grade III-IV (Toxicity Criteria of the South West Oncology Group, 1992) - with a negative benefit/risk ratio
* severe renal disease (Creatinin Clearance < 30 ml/min)
* severe liver disease (AST or ALT > 5-times normal)
* coexisting, malignant, systemic diseases

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2002-09

CONTACTS AND LOCATIONS:
Locations (24):
- Austria (3):
  - Center Innsbruck, Innsbruck, Tyrol
  - Center AKH, Vienna, Vienna
  - Center Hanusch, Vienna, Vienna
- Czechia (3):
  - Center Brno, Brno
  - Center Olomouc, Olomouc
  - Center Praha, Prague
- Center Paris, Paris, Clichy Cedex, France
- Germany (5):
  - Center Munich, Munich, Bavaria
  - Center Berlin, Berlin
  - Center Halle, Halle
  - Center Saarbrücken, Saarbrücken
  - Center Ulm, Ulm
- Center Budapest, Budapest, Hungary
- Italy (2):
  - Center Modena, Modena
  - Center Pavia, Pavia
- Center Vilnius, Vilnius, Lithuania
- Poland (6):
  - Center Gdansk, Gdansk
  - Center Katowice, Katowice
  - Center Krakow, Krakow
  - Center Lodz, Lodz
  - Center Lublin, Lublin
  - Center Warszawa, Warsaw
- Center Singapore, Singapore, Singapore
- Center Ljubljana, Ljubljana, Slovenia

REFERENCES:
- [Derived] Gisslinger H, Gotic M, Holowiecki J, Penka M, Thiele J, Kvasnicka HM, Kralovics R, Petrides PE; ANAHYDRET Study Group. Anagrelide compared with hydroxyurea in WHO-classified essential thrombocythemia: the ANAHYDRET Study, a randomized controlled trial. Blood. 2013 Mar 7;121(10):1720-8. doi: 10.1182/blood-2012-07-443770. Epub 2013 Jan 11. PMID 23315161